CLINICAL TRIAL: NCT04014595
Title: The Evaluation of a Strategy to PREPARE Severely CALCified Coronary Lesions With a Combination Of Rotational Atherectomy and Modified BallOons Trial (PREPARE-CALC- COMBO)
Brief Title: PREPARE-CALC-COMBO: Severely Calcified Coronary Lesions Prepared With Rotational Atherectomy and Modified Balloons
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SK 110 -- 168/11
Record Dates: First submitted 2019-06-28; First posted 2019-07-10 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
Keywords: Calcified coronary lesions
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Rotational atherectomy + Cutting Balloon: Rotational atherectomy in combination with cutting balloon in severely calcified coronary lesions
  Interventions: Procedure: Rotational atherectomy in combination with cutting balloon

INTERVENTIONS:
Procedure: Rotational atherectomy in combination with cutting balloon — Treatment of severely calcified coronary lesion using rotational atherectomy followed by balloon angioplasty using a cutting balloon and Implantation of the hybrid sirolimus-eluting stent.

SUMMARY:
A prospective single-arm trial of rotational atherectomy in combination with cutting balloon in severely calcified coronary lesions.

DETAILED DESCRIPTION:
A prospective single-arm trial to evaluate the acute and long term efficacy of a combined strategy of lesion preparation with rotational atherectomy followed by cutting balloon and by hybrid sirolimus-eluting stent implantation in an angiographically well-defined group of patients with severely calcified coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria

1. Age above 18 years and consentable
2. Angiographically proven coronary artery disease
3. Anginal symptoms and/or reproducible ischemia in the target area by ECG, functional stress testing or fractional flow reserve
4. Written informed consent

Angiographic inclusion criteria

1. De-novo lesion in a native coronary artery
2. Target reference vessel diameter between 2.25 and 4.0 mm by visual estimation
3. Luminal diameter reduction of 50-100% by visual estimation
4. Severe calcification of the target lesion (for definition see appendix)

Exclusion Criteria:

Clinical exclusion criteria

1. Myocardial infarction (within 1 week)
2. Decompensated heart failure
3. Limited long term prognosis due to other conditions

Angiographic exclusion criteria

1. Target lesion is in a coronary artery bypass graft
2. Target lesion is an in-stent restenosis
3. Target vessel thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease subjected to percutaneous revascularization of the native coronary arteries and fullfilling all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: Numerical in-stent acute lumen gain in mm | At the end of the index procedure
  The main angiographic endpoint will be in-stent acute lumen gain defined as minimal lumen diameter (MLD) in stent at the end of the index procedure minus baseline MLD.
Co-primary OCT endpoint: Ratio of stent expansion index (SEI) | At the end of the index procedure
  The main OCT endpoint will be stent expansion index (SEI), defined as minimum stent area divided by mean reference area in optical coherence tomography (OCT) quantitative analysis at the end of the index procedure

SECONDARY OUTCOMES:
Numerical in-stent late lumen loss at 9 month follow-up angiography in mm | 9 months follow-up
  In-stent late lumen loss at 9 month follow-up angiography defined as the difference between the postprocedure in-stent minimal lumen diameter (MLD)and the in-stent MLD at 9-month followup angiography will be adopted as a co-primary endpoint.
Rate of angiographic success in percent | Peri-procedural
  'Angiographic Success' defined as successful stent delivery and expansion with attainment of < 20% in-stent residual stenosis of the target lesion in the presence of TIMI 3 flow.
Rate of strategy success in percent | Peri-procedural
  'Strategy Success' defined as successful stent delivery and expansion with attainment of < 20% in-stent residual stenosis of the target lesion in the presence of TIMI 3 flow without stent failure.
Rate of target vessel failure in percent | 9 months, 1 and 2 years follow-up
  Target vessel failure (TVF) defined as a composite of cardiac death, target vessel related myocardial infarction and clinically driven target vessel revascularization at 9 months, 1 and 2 years.
Rate of in-segment binary restenosis at 9 months in percent | 9 months follow-up
  In-segment binary restenosis at 9 months
Rate of stent thrombosis in percent | 9 months, 1 and 2 years follow-up and final 5 years follow-up
  Stent thrombosis
Rate of peri-procedural myocardial infarction in percent | Peri-procedural
  Peri-procedural myocardial infarction
Rate of vessel perforation in percent | Peri-procedural
  Rate of vessel perforation
Numerical procedural duration in min | Peri-procedural
  Procedural duration
Numerical contrast dye amount in ml | Peri-procedural
  Procedural contrast dye amount

OTHER OUTCOMES:
Ratio of OCT-measured stent excentricity index | Intra-procedural
  Defined as the ratio of minimal lumen diameter and the maximal lumen diameter per cross section at the end of index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gert Richardt, Prof., Study Chair — Herzzentrum Segeberger Kliniken GmbH
Locations (1):
- Herzzentrum Segeberger Kliniken GmbH, Bad Segeberg, Germany